CLINICAL TRIAL: NCT06520657
Title: Addressing Social Determinants of Health in Child Obesity Treatment Using Community Health Workers: the Role of Parental Bandwidth in Treatment Effectiveness
Brief Title: Addressing Social Determinants of Health in Child Obesity Treatment Using Community Health Workers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Community Health Council of Wyandotte County (Unknown); University of Kansas Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Helena Laroche, MD, Physician, MD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002819; 1R01DK139363-01 (NIH)
Record Dates: First submitted 2024-07-02; First posted 2024-07-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Child Obesity; Social Determinants of Health
Keywords: Community Health Workers; Randomized trial; Pilot Study; Child Obesity Treatment; Executive function
MeSH Terms: conditions — Pediatric Obesity | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: 60 Families (2 participants in each- parent and child) will be randomized to community health worker intervention or standard social risk factor (SRF) referral for the first 3 months and then 3-6 months both groups will do the same child obesity intervention then 6-12 months both will receive no intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHW plus child weight management intervention (Experimental): Participants in this arm will work with a community health worker for three months to address social risk factors (negative social determinants of health) prior to beginning a child weight management group treatment.
  Interventions: Other: Community Health Worker; Behavioral: Child weight management intervention; Other: Standard of Care referral to resources
- Child weight management intervention only (Active Comparator): Participants in this arm will receive the standard of care which includes a one-time referral to community resources to meet their social needs. At three months they also begin the same child weight management group treatment as the experimental group.
  Interventions: Behavioral: Child weight management intervention; Other: Standard of Care referral to resources

INTERVENTIONS:
Other: Community Health Worker — Participants are screened for social determinants of health and work with a community health worker for three months to connect them with community and government services to address their family's needs.
  Arms: CHW plus child weight management intervention
Behavioral: Child weight management intervention — This is a 12-week family-based behavioral group intervention to address childhood overweight and obesity.
Other: Standard of Care referral to resources — One-time referral to resources based on need that families can access independently either by providing electronic referral to or providing written contact information for a community resource.

SUMMARY:
The goal of this small pilot study is to test the feasibility of combining a three-month intervention of working with a community health worker (CHW) to address social risk factors for patients prior to beginning a group weight management program for childhood obesity -- Promoting Health in Teens and Kids (PHIT Kids)

ELIGIBILITY:
Inclusion Criteria:

* Family must have one major social risk factor on the Protocol for Responding to & Assessing Patients' Assets, Risks & Experiences (PRAPARE) of the 14 modifiable risk factors
* Child aged 8 through 12 years of age
* Child with BMI% at 85th percentile or higher and less than the 120% of the 95th percentile (overweight or class 1 obesity)
* Child must live with parent/guardian at least 5 out of the 7 days on average (70% of the time)
* Child and parent able to speak English

Exclusion Criteria:

* Child on medications known to cause ongoing weight gain (e.g., atypical anti-psychotics, chronic prednisone, insulin)
* Child on other medications know to affect weight if dose and BMI z-score has not been stable for 3 months.
* Diabetes or other disease that has a significant effect on diet, physical activity, or ability to take part in trial activities besides obesity (does not included treated or mild depression or anxiety, limited food allergies or mild physical activity limitations)
* For parents: new MI, stroke or cancer diagnosis (excluding localized skin cancers) in past 6 months, history of bariatric surgery within the past 3 years, pregnancy in last 6 months or planned within 1 year
* Child or parent has significant developmental or cognitive impairments or other significant medical issue that would interfere with ability to participate or complete assessment
* Parent or child has significant physical limitation
* Parent/child planning to move to from Children's Mercy Kansas City (CMKC) service area

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment Rate | 1 year
  Number of participants enrolled (consented) per month
Retention | 6 months
  Attendance at 6 month data assessment
Satisfaction with Community Health Worker (CHW) | 3 months
  A 15-item scale asks about quality of interactions and satisfaction with their CHW. Scores range from 15 to 60, with higher scores indicating increased satisfaction.
Satisfaction with PHIT Kids - Parent | 6 months
  A single 10-point Likert scale satisfaction rating about the group weight management intervention. Scores range from 1-10 with higher scores indicating increased satisfaction.
Child Body Mass Index (BMI) Z-Score | Change in BMI Z-score over a 6 month time period in the child with obesity or overweight
  6 months
Inhibitory Control and Attention | 3 months
  The Flanker Inhibitory and Control Attention Test (Flanker) measures accuracy and reaction time to produce a combined score ranging from 0-10 with higher scores indicating better inhibitory control and attention.
Working Memory | 3 months
  The List Sorting Working Memory Test asks participants to recall a list of foods and animals in order from smallest to largest. Correct responses range from 0-26, and are then converted to nationally normed standard scores ranging from 59-140, with higher scores indicating better working memory.
Cognitive Flexibility | 3 months
  The Dimensional Change Card Sort Test (DCCS) measures accuracy and reaction time to produce a combined score ranging from 0-10 with higher scores indicating better cognitive flexibility.
Parent Cognitive Capacity | 3 months
  The Raven's 2 Progressive Matrices- Digital Short Form (Raven's 2) tests fluid intelligence by asking participants to identify missing pieces in visual geometric patterns of up to 24 progressively more difficult trials. The total number correct is converted into Standard Scores, which will be compared to a participant's other scores over the course of the study. Standard scores range from 59-140 with higher scores indicating increased cognitive capacity.

SECONDARY OUTCOMES:
PHIT Kids attendance | 6 months
  percent of PHIT Kids sessions attended
Percentage of needs met or partially met | 3 months
  At 3 months, participants will review each need identified at baseline and report if they received "All the help I needed," "Most of the help I needed," "A little of the help I needed," or "None of the help I needed." The total number of needs that were at least partially met ("a little", "most" or "all") or that were fully met ("all") will be divided by the total number of needs at baseline
Enrollment in at least one new resource | 3 months
  Yes/No. Family has accessed at 3 months at least one new community or government resource since baseline. Participants will review a list of resources potentially offered to CHW clients and respond whether they currently receive this resource at baseline and 3 months
Number of key measures completed | 6 months
  Number of the following measures completed - outcome measures (child BMI-z, parent weight, MVPA (actigraph; at least 4 days), dietary measures (3 recalls)), bandwidth measures (executive functions measures and Raven matrices) and self-efficacy.
Parent Weight | 6 months and 12 months
  Change in parent weight at 6 month and 12 months
Child Moderate to Vigorous Physical Activity (MVPA) | 6 months and 12 months
  Minutes per week in moderate to vigourous physical activity as measure by an Actigraph waist accelerometer worn by the child. Also percent of time in MVPA
Child Dietary Intake | 6 months and 12 months
  Three 24 hour recalls completed by parent using the he Automated Self-Administered 24-hour Dietary Assessment Tool (ASA 24) computer program - used to calculate fruit and vegetable (FV) servings, sugar sweetened beverages, and number of high fat/high sugar foods (foods with >7g of fat and/or 12g of sugar)
Self-Efficacy | 6 months
  10-item, 5-point Likert scale. Measured by the General Self-Efficacy Scale in the NIH Toolbox. This scale assesses an individual's perceived ability to cope with stressful situations. Scores range from 10 to 50 with higher scores indicating higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Laroche, MD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided